CLINICAL TRIAL: NCT04971382
Title: Alveolar Ridge Augmentation With Curcumin Combined With Xenograft After Piezoelectric Alveolar Ridge Splitting Surgery (A Randomized Controlled Clinical Trial)
Brief Title: Alveolar Ridge Augmentation With Curcumin Combined With Xenograft
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasmine Gamal, Ass.lecturer of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMD2021-3-
Record Dates: First submitted 2021-07-05; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Horizontal Alveolar Bone Loss
Keywords: curcumin; xenograft; Piezoelectric; Alveolar Ridge Splitting
MeSH Terms: interventions — Curcumin; turmeric extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- curcumin combined with particulate xenograft. (Experimental): Curcumin will be used in combination with xenograft after ridge splitting surgery
  Curcumin is widely used in medicine due to medicinal properties, cost-effectiveness, and simple extraction from a turmeric plant that grows in different regions in the world. Recent evidences have shown that curcumin possesses multiple biological activities and pharmacological properties including anti-inflammation , antioxidation , anticancer , antimicrobial , and free radical scavenger effects
  Interventions: Drug: Curcumin
- alveolar ridge splitting with use of particulate xenograft alone. (Active Comparator): xenograft will be used alone after ridge splitting
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Curcumin — Curcumin (1,7-bis(4-hydroxy-3-methoxyphenyl)-1,6-heptadiene-3,5-dione) or diferuloylmethane is an important bioactive constituent and hydrophobic polyphenol that isolated from the rhizome of the turmeric plant (Curcuma longa) . Curcumin will be used in combination with xenograft after ridge splitting surgery
  Other Names: Curcumin (Curcuma longa)

SUMMARY:
A study was performed to investigate the effect of curcumin on the osteogenic differentiation of human periodontal ligament stem cells (hPDLSCs) and its underlying potential mechanism. The Results was that Curcumin at an appropriate concentration had no cytotoxicity and could promote osteogenic differentiation of the hPDLSCs

DETAILED DESCRIPTION:
Patients will be selected from the outpatient clinic of Oral Medicine, Periodontology and Oral diagnosis Department, Faculty of Dentistry, Ain Shams University. The purpose of the study will be explained to all patients and an informed consent will be signed before the conduction of the study .The faculty research ethics committee will review the proposal.

The study will be conducted in the form of Patient Intervention Comparative Outcome (PICO) question (Patient "P", Intervention "I", Comparative "C", Outcome "O"). (Stone 2002) "P": Patient in the study will have enough alveolar ridge height ,suffering from missing from 1 to 3 upper maxillary anterior and /or premolar with insufficient alveolar ridge buccolingual (BL) width that interfere with conventional straight forward implant placement. The minimum BL width included in the study will be 4 mm. "I": Ridge splitting with interposition grafting with curcumin and particulate xenograft grafting. "C":Alveolar ridge splitting with interposition grafting with use of particulate xenograft alone without curcumin . "O":Clinical and radiographic outcome.

ELIGIBILITY:
Inclusion Criteria:

* Male and female with age range 25-45 years.
* Patient with enough alveolar ridge height, suffering from missing single or multiple maxillary anterior and /or premolar with insufficient alveolar ridge buccolingual (BL) width that interfere with conventional straight forward implant placement. The minimum BL width included in the study will be 4-5 mm to facilitate ridge splitting and expansion.
* Systemically free from any diseases as evidenced by Burket's oral medicine health history questionnaire.
* Patient available during follow up periods.

Exclusion Criteria:

* Smokers.
* Pregnant and breast feeding females.
* Patient unwilling to comply to oral hygienic instructions.
* Patients under any medication or medical condition that affect the bone quality.
* Vulnerable groups. (e.g decisions impaired individual).

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
clinical outcome | change from baseline at 6 months
  Assessment the gain in alveolar ridge buccolingual width

SECONDARY OUTCOMES:
stability | "through study completion, an average of 1 year
  Assessment of the primary implant stability Quotient in the regenerated bone

CONTACTS AND LOCATIONS:
Overall Officials: Hala A Abuelela, professor, Study Director — faculty of dentistry . Ain Shams University
Locations (1):
- faculty of dentistry Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No